CLINICAL TRIAL: NCT07317336
Title: I-SLEPT: Integrated Sleep and Life Engagement Program for Transitions
Acronym: I-SLEPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRD9-010-25M; 1IK2RD000347-01A1 (Other Grant/Funding Number: RRDT)
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Sleep; Participation
Keywords: sleep; participation; rehabilitation; transitions of care; physical function

STUDY DESIGN:
Intervention Model Description: Assess for feasibility and clinically significant results of I-SLEPT in a proof-of-concept, single-arm trail in Veterans (Enrollment Target; N = 60) age 50 years and older who were recently discharged from VA Boston Subacute Rehabilitation to home. Targeting 40 completers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- I-SLEPT (Experimental): Veterans in Aim 3 will complete I-SLEPT, a 4-week telehealth intervention, delivered by a licensed clinical psychologist. Sessions will take place once a week for 60 minutes primarily using VA Video Connect. Sessions will include components focused on 1) promoting sleep health through education and habits and 2) increase engagement in meaningful activities.
  Interventions: Behavioral: I-SLEPT

INTERVENTIONS:
Behavioral: I-SLEPT — Veterans in Aim 3 will complete I-SLEPT, a 4-week telehealth intervention, delivered by a licensed clinical psychologist. Sessions will take place once a week for 60 minutes primarily using VA Video Connect. Sessions will include components focused on 1) promoting sleep health through education and habits and 2) increase engagement in meaningful activities.

SUMMARY:
Sleep is essential to functional recovery in rehabilitation settings; however, sleep is likely to be disrupted during rehabilitation admissions. Adverse effects of these disruptions do not subside after discharge, leading to additional consequences such as poor physical function. Veterans are particularly impacted by poor sleep and medical complexities that can lead to injuries requiring rehabilitative care to support their recovery. This may be more apparent in older Veteran populations. After discharge, Veterans must re-acclimate to their home environment while facing potential changes in their sleep, life engagement (e.g., pleasant activities, physical function), and health. This study will create the I-SLEPT (Integrated Sleep and Life Engagement Program for Transitions) intervention, which will support Veterans by stabilizing their sleep and by maximizing participation in meaningful activities during a critical and vulnerable period of recovery.

DETAILED DESCRIPTION:
This project will create I-SLEPT (Integrated Sleep and Life Engagement Program for Transitions), a novel intervention to enhance sleep health and life engagement during the transition period following discharge from VA subacute rehabilitation. The development of I-SLEPT will be informed by both Veterans and experts. Including the Veteran perspective is essential to reflect Veterans' choice, ensure access to timely care, and prioritize effective care solutions to improve Veterans' health and well-being. Veterans are more likely to report poor sleep and medical complexities than non-Veterans which may further complicate their readjustment to their home environment after discharge. The proposed study is a single arm clinical trial. Veterans aged 50+ discharged home from the subacute rehabilitation units at VA Boston's Community Living Center will be recruited to complete surveys and interviews informing I-SLEPT creation (Aim 1; N=20), complete a preliminary trial (Aim 2; N=5) or complete a single-arm Proof-of-Concept trial (Aim 3; N=40). Veterans participating in Aims 2 or 3 will complete assessments of sleep health and life engagement, as well as acceptability measures. Results may also inform future work adapting this intervention to other transitional phases (e.g., discharge from acute hospitalization), support Veterans across the lifespan, and support intervention implementation by staff from multiple disciplines and specialties, including nursing, social work, physical therapy, occupational therapy, and Veteran peer specialists.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to and discharged from VA Boston Community Living Center subacute rehabilitation
* English-speaking
* Discharged to a home setting
* Has capacity and does not have severe cognitive impairment
* Obtains a score >= 8 on the Brief Interview for Mental Status (BIMS)
* Endorses at least 2 items as "Rarely/Never" or "Sometimes" on the RuSATED measure AND/OR endorses they are achieving their goals at a "much worse" or "a little worse" level on the What Matters Most Tool.

Exclusion Criteria:

* Discharged from Long-Term Care, Hospice and Palliative Care, or Spinal Cord Injury bed specialty
* Moderate to severe dementia diagnosis, delirium, or active psychosis
* Healthcare proxy is activated in electronic health record
* A diagnosis of a disorder of hypersomnolence, non-REM parasomnia, or Nightmare Disorder as indicated in electronic health record
* High acute risk for suicide

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04-03 (Estimated); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
RuSATED | Baseline, Endpoint (30 day), 3 Month
  A brief 6-item measure encompassing the dimensions of sleep health: Regularity, Satisfaction, Alertness, Timing, Efficiency, and Duration. Scores range from 0 to 12 with higher total scores suggesting better sleep health. Items are rated on a 3-point scale from 0 to 2 (with 0 = Rarely/Never; 1 = Sometimes; and 2 = Usually/Always).
What Matters Most (WMM) Tool | Baseline, Endpoint (30 day), 3 Month
  A one-page brief tool presenting 3 domains (Staying Independent, Enjoying Life, and Connecting), each containing a list of 9 items with the option of adding a 10th item of their own. Veterans will be asked to identify up to 3 items within each domain that matters most to them. After up to 9 items total have been identified, Veterans will be asked to "pick the most important thing" and describe what this would look like for them "day to day or week to week." Veterans will be encouraged to pick up to 3 things that matter most above all. Finally, Veterans are asked to rate how well they are achieving their life engagement goals and what matters most to them, employing a 5-point Likert-style goal attainment scale (+2 = much better than expected; +1 = a little better than expected; 0 = as expected; -1 = a little worse than expected; -2 = much worse than expected). A score of 0-2 indicate satisfactory goal attainment in the ar
Acceptability of Intervention Measure (AIM) | Endpoint (30 day)
  A 4-item measure that assess acceptability, defined here as the perception that I-SLEPT is acceptable, palatable, or satisfactory.
Feasibility of Intervention Measure (FIM) | Endpoint (30 day)
  A 4-item measure that assesses feasibility defined here as the extent to which the session material can be successfully used - defined as from the Veteran's perspective of applying what is learned after the session.

SECONDARY OUTCOMES:
Intervention Appropriateness Measure (IAM) | Endpoint (30 day)
  A 4-item measure that assesses appropriateness, defined here as the Veteran's perspective on the perceived fit, relevance, or compatibility of session material to the Veteran's sleep health and life engagement concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Julia T Boyle, PsyD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No